CLINICAL TRIAL: NCT05868733
Title: A Phase 2 Randomized, Double-Blinded, Placebo-Controlled Clinical Trial to Evaluate the Safety, Tolerability, and Immunogenicity of rVSV∆G-LASV-GPC Vaccine in Adults and Children Residing in West Africa
Brief Title: A Lassa Fever Vaccine Trial in Adults and Children Residing in West Africa
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: International AIDS Vaccine Initiative (Network)
Collaborators: Coalition for Epidemic Preparedness Innovations (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Prevention
Other Study IDs: IAVI C105
Record Dates: First submitted 2023-05-08; First posted 2023-05-22 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Lassa Fever
MeSH Terms: conditions — Lassa Fever

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Study staff and participants will be blinded in terms of active product versus placebo.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (10):
- Cohort 1A (Experimental): Healthy Adults, 18-70yrs
  Interventions: Drug: Day 1 Lower Dose (2×106 pfu); Drug: Placebo
- Cohort 2A (Experimental): HIV-infected Adults, 18-50yrs
  Interventions: Drug: Day 1 Lower Dose (2×106 pfu); Drug: Placebo
- Cohort 3A (Experimental): Adolescents, 12 17yrs
  Interventions: Drug: Day 1 Lower Dose (2×106 pfu); Drug: Placebo
- Cohort 4A (Experimental): Children, 6-11yrs
  Interventions: Drug: Day 1 Lower Dose (2×106 pfu); Drug: Placebo
- Cohort 5A (Experimental): Children, 18mos-5yrs
  Interventions: Drug: Day 1 Lower Dose (2×106 pfu); Drug: Placebo
- Cohort 1B (Experimental): Healthy Adults, 18-70yrs
  Interventions: Drug: Day 1 Higher Dose (1×107 pfu); Drug: Placebo
- Cohort 2B (Experimental): HIV-infected Adults,18-50yrs
  Interventions: Drug: Day 1 Higher Dose (1×107 pfu); Drug: Placebo
- Cohort 3B (Experimental): Adolescents, 12 17yrs
  Interventions: Drug: Day 1 Higher Dose (1×107 pfu); Drug: Placebo
- Cohort 4B (Experimental): Children, 6-11yrs
  Interventions: Drug: Day 1 Higher Dose (1×107 pfu); Drug: Placebo
- Cohort 5B (Experimental): Children, 18mos-5yrs
  Interventions: Drug: Day 1 Higher Dose (1×107 pfu); Drug: Placebo

INTERVENTIONS:
Drug: Day 1 Lower Dose (2×106 pfu) — rVSV∆G-LASV-GPC
  Arms: Cohort 1A; Cohort 2A; Cohort 3A; Cohort 4A; Cohort 5A
Drug: Day 1 Higher Dose (1×107 pfu) — rVSV∆G-LASV-GPC
  Arms: Cohort 1B; Cohort 2B; Cohort 3B; Cohort 4B; Cohort 5B
Drug: Placebo — Placebo

SUMMARY:
A Phase 2 Randomized, Double-Blinded, Placebo-Controlled Clinical Trial to Evaluate the Safety, Tolerability, and Immunogenicity of rVSV∆G-LASV-GPC Vaccine in Adults and Children Residing in West Africa

DETAILED DESCRIPTION:
rVSVΔG-LASV-GPC is a candidate vaccine that has been shown to be safe and protects against LF disease in animals. The vaccine was studied studied in a Phase 1 trial and has been well tolerated and immunogenic. This Phase 2 trial will add to data from the Phase 1 trial to establish a broader profile of safety and immunogenicity in adults and expand the population to include a subset of adults with HIV infection as well as older adults and healthy children, in preparation for an efficacy trial in West Africa. Primary Objective: • To evaluate the safety and tolerability of rVSVΔG-LASV-GPC vaccine at 2 different dosage levels in adults, including PLWH, and in children Secondary Objectives: • To determine binding LASV-GPC-specific antibody responses induced by rVSVΔG-LASV-GPC vaccine • To determine neutralizing LASV-GPC-specific antibody responses induced by rVSVΔG-LASV-GPC vaccine in a subset of participants in each group • To evaluate the magnitude and duration of the rVSVΔG-LASV-GPC vaccine viremia in plasma in a subset of participants. • To evaluate the magnitude and duration of the rVSVΔG-LASV-GPC vaccine shedding in saliva and urine, and possibly semen and cervicovaginal fluid, in a subset of participants Exploratory Objective • To explore the characteristics of the immune responses induced by rVSVΔG-LASV-GPC vaccine in a subset of participants

ELIGIBILITY:
Inclusion Criteria:

* Adults, adolescents, and children in good general health as assessed by medical history and physical examination (group-specific criteria apply).
* At least 18 months old on the day of screening and not more than 70 years old on the day of vaccination (group-specific criteria apply).
* Participant or parent/guardian willing to comply with the requirements of the protocol and available for follow-up for the planned duration of the study.
* In the opinion of the Principal Investigator (PI) or designee and based on Assessment of Informed Consent Understanding (AOU), participant or parent/guardian has understood the information provided and potential impact and/or risks linked to administration and participation in the trial; written informed consent will be obtained before any study-related procedures are performed. Children old enough to understand the procedures will be asked to assent, in addition to parent/guardian consent, in accordance with local requirements.
* Willing to undergo HIV testing, risk reduction counselling, and receive HIV test results (group-specific timepoints apply).
* All participants of child-bearing potential engaging in sexual activity that could lead to pregnancy must commit to use an effective hormonal contraception or intrauterine device beginning 2 weeks prior and extending for 4 months following receipt of vaccine/placebo. Study sites will choose which methods are most appropriate for their population and this will be specified in the Informed Consent Document (ICD).
* All sexually active participants must consistently use male or female condoms with all sexual partners for 4 months following IP administration.
* All participants who are not engaging in sexual activity that could lead to pregnancy at screening must agree to utilize an effective method of contraception if they begin engaging in sexual activity that could lead to pregnancy, as outlined above.
* All participants of childbearing potential must be willing to undergo a pregnancy test at time points indicated in the SOA.
* Willing to forgo donation of blood or any other tissues for transfusion or transplantation, from screening onward throughout the course of the study.

Additional Inclusion Criteria For HIV-Infected Participants

* Adults who are HIV-infected must meet the following additional inclusion criteria:
* Participant must be aged at least 18 years old on the day of screening and not more than 50 years old on the day of vaccination.
* Participant must have documented HIV-1 or HIV-2 infection for at least 6 months prior to screening.
* Participant must be on a stable (at least 6 months) regimen of Highly Active Antiretroviral Therapy (HAART), as defined as potent anti-HIV treatment including a combination of antiretroviral agents (pre- or post-exposure prophylaxis does not count as HAART).
* Participant entering the study should have a screening viral load <50 copies/ml.
* Participant must be willing to continue their HAART and HIV care follow up throughout the study as directed by their regular caregiver and be willing to give access to records of their ongoing care.
* Participant must be in an otherwise reasonably good medical condition (absence of acquired immunodeficiency syndrome [AIDS]-defining illnesses or clinically significant disease), diagnosed based on physical examination, medical history, and the investigator's clinical judgment.

Additional Inclusion Criteria for Pediatric Participants

* Each potential pediatric study participant must meet all of the following additional criteria to be enrolled in the study:
* Parent(s)/legal guardian must have signed an ICD indicating that they understand the purpose and procedures required for the study, are willing/able to adhere to the study requirements and are willing for their child to participate in the study. Assent must be obtained from adolescents and children in accordance with local regulations and practice. Parent(s)/legal guardian must pass the AOU.
* Participant's age on the day of vaccination is within one of the 3 age strata in the study: 12-17 years, 6-11 years, or 18 months -5 years.
* Participant must be healthy in the investigator's clinical judgment (and the parent(s)/legal guardian's judgment) based on medical history, physical examination and vital signs performed at screening.
* A female adolescent who is of childbearing potential must comply with requirements for contraception.
* Adolescents who are sexually active must comply with requirement for use of condoms for 4 months after vaccination.
* Participant has received all routine immunizations appropriate for their age as reported by the parent(s)/legal guardian, according to local routine vaccination schedules. Participants are allowed to catch up on routine immunizations if needed or as part of national immunization campaigns. However, Exclusion Criteria #9 will apply.

Exclusion Criteria:

* Confirmed HIV-1 or HIV-2 infection (except as outlined for Group 2)
* Any clinically relevant abnormality on history or examination including history of immunodeficiency (except for Group 2) or autoimmune disease; use of corticosteroids, immunosuppressive, anticancer, or other medications considered significant by the Investigator within the previous 6 months. The following exceptions are permitted and will not preclude study participation: use of corticosteroid nasal spray for rhinitis, topical corticosteroids for an acute uncomplicated dermatitis; or a short course (duration of 10 days or less, or a single injection) of corticosteroid for a non-chronic condition (based on Investigator clinical judgment) at least 2 weeks prior to enrollment in this study.
* Any clinically significant chronic medical condition that, in the opinion of the Investigator, makes the participant unsuitable for participation in the study (except for HIV in Group 2). Note: Participants aged >50years with the following chronic but controlled conditions may be enrolled:
* Hypertension with systolic ≤150 mmHg and/or diastolic ≤90 mmHg; (regardless of treatment status)
* Diabetes mellitus with a HbA1C <10% and /or with type 2 diabetes mellitus on stable medication for at least 2 months prior to enrollment.
* Pregnant or lactating.
* Bleeding disorder that was diagnosed by a physician (eg, factor deficiency, coagulopathy, or platelet disorder that requires special precautions). Note: A participant who states that he or she has easy bruising or bleeding but does not have a formal diagnosis and has intramuscular (IM) injections and blood draws without any adverse experience is eligible.
* Infectious disease: chronic active hepatitis B infection (HBsAg-positive), current hepatitis C infection, prior clinical diagnosis of Lassa Fever disease (LF) or Ebola virus disease (EVD) by medical history, active syphilis (positive screening and confirmatory tests unless adequately treated), positive viral detection test for SARS-CoV-2. Note: COVID-19 screening is not applicable for Group 5.
* History of splenectomy or functional asplenia.
* Any of the following abnormal laboratory parameters listed below:
* Hematology
* Absolute Neutrophil Count (ANC): ≤1,000 cells/mm3 or ≤ 1.0 × 109 cells/L
* Absolute Lymphocyte Count (ALC): ≤650 cells/mm3 or ≤ 0.65 × 109 cells/L
* Hemoglobin: <9.5 g/dl in females; <11.0 g/dl in males; <10 g/dl in children <11 years of age
* Platelets <100,000 cells/mm3
* Chemistry
* Creatinine >1.1 x upper limit of normal (ULN) (Note: For participants aged >50 years clinically insignificant renal insufficiency defined as creatinine ≤1.3 x ULN is allowed)
* Alanine transaminase (ALT) >1.25 x ULN
* Aspartate transaminase (AST) >1.25 x ULN
* Urinalysis (not applicable for group 5)
* Clinically significant abnormal dipstick confirmed by repeat dipstick on new specimen or by microscopy
* Protein = 1+ or more
* Blood = 2+ or more (not due to menses) (Urinalysis may be collected within the following 2 weeks if menses interfere)
* Receipt of any vaccine within the previous 28 days or planned receipt within 28 days after vaccination with IP. Participation may be delayed until this criterion can be fulfilled. Note: prior receipt of VSV-vectored vaccines such as VSV-ZEBOV will be documented but is not an exclusion criterion.
* Prior receipt of another investigational Lassa vaccine candidate. Note: receipt of placebo in a previous LF vaccine trial will not exclude a participant from participation if documentation is available and the Medical Monitor gives approval.
* Receipt of blood transfusion or blood-derived products within the previous 3 months.
* Participation in another clinical trial or observational study currently, within the previous 3 months, or expected participation during this study, unless Medical Monitor approves.
* History of severe local or systemic reactogenicity to any vaccine (eg, anaphylaxis, respiratory difficulties, angioedema, injection site necrosis, or ulceration).
* Psychiatric condition or substance abuse that compromises safety of the participant and precludes compliance with the protocol. Specifically excluded are persons with psychoses in the last 3 years prior to screening, ongoing risk for suicide, or history of suicide attempt or gesture in the last 3 years prior to screening.
* Seizure disorder: A participant who has had a seizure in the last 3 years prior to screening or has been on any medication to control or prevent seizures for the last 3 years is excluded. Group 5: History of febrile seizures is an exclusion criterion.
* A history of malignancy in the past 5 years (prior to screening) or ongoing malignancy (a history of a completely excised malignancy that is considered cured is not an exclusion).
* Active, serious infections requiring parenteral antibiotic, antiviral, antiparasitic or antifungal therapy within 30 days prior to enrollment (except HAART treatment in Group 2). Asymptomatic malaria infection at study entry will be assessed retrospectively and will not be a basis for exclusion.
* Group specific weight for height restrictions as indicated below:
* Groups 1 and 2: Obesity as defined by Body mass index (BMI) ≥35.
* Group 3: Obesity as defined by weight for height 2 standard deviation (SD) from median according to WHO growth charts or underweight as defined by weight for height or weight for length ≤-2 SD from median according to WHO growth charts
* Groups 4 and 5: Underweight as defined by weight for height or weight for length ≤ 2 SD from median according to WHO growth charts (see APPENDIX C) and/or weighing <10kg.
* Group specific hearing thresholds or otoacoustic emission (OAE) results at 0.5-4KHz as indicated below:
* Moderate or greater hearing impairment defined as 35dB in any frequency in either ear as revealed via the audiometry exam for Groups 1 and 2.
* Mild or greater hearing impairment defined as ≥20dB in any frequency in either ear as revealed via the audiometry exam for adolescents and children aged >7years.

For children 7 years of age and younger (or unable to follow pure tone audiometry procedure) "refer" test results as determined by OAE.

* Otorrhea within the past 90 days, sudden or rapid hearing loss within the past 90 days, acute or chronic dizziness, otalgia (external ear otalgia is not an exclusion)
* Clinically relevant abnormal otoscopy, that in the opinion of the investigator, may interfere with hearing. (Participants with conditions that can be treated prior to enrolment such as cerumen obstruction are not excluded)
* History of acute or chronic or severe neurologic condition (eg, diagnosis of Guillain-Barré syndrome, epilepsy, Bell's palsy, meningitis, or disease with any focal neurologic deficits).
* Current of past significant risk factors for hearing loss (eg, occupational exposure to loud noise or medical illness) that, in the opinion of the investigator, may interfere with the detection of changes in hearing during the study.
* History of any condition associated with sensorineural hearing loss that, in the opinion of the investigator, may cause changes in hearing during the study (eg, occupational exposure to loud noise or medical illness).
* If, in the opinion of the PI, it is not in the best interest of the participant to participate in the study.

Ages: 18 Months to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 612 (Estimated)
Dates: Start 2024-03-06 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of rVSV∆G-LASV-GPC vaccine at 2 different dosage levels in adults, including PLWH, and in children | 14 days
  Proportion of participants with Grade 3 or higher reactogenicity, ie, solicited AEs, within 14 days after IP administration
To evaluate the safety and tolerability of rVSV∆G-LASV-GPC vaccine at 2 different dosage levels in adults, including PLWH, and in children | 28 days
  Proportion of participants with IP-related Grade 2 or higher unsolicited AEs, including safety laboratory parameters, within 28 days of IP administration
To evaluate the safety and tolerability of rVSV∆G-LASV-GPC vaccine at 2 different dosage levels in adults, including PLWH, and in children | 28 days
  Proportion of participants with any Grade 2 or higher unsolicited AEs, including safety laboratory parameters, within 28 days of IP administration
To evaluate the safety and tolerability of rVSV∆G-LASV-GPC vaccine at 2 different dosage levels in adults, including PLWH, and in children | 7 months
  Proportion of participants with IP-related SAEs throughout the study period
To evaluate the safety and tolerability of rVSV∆G-LASV-GPC vaccine at 2 different dosage levels in adults, including PLWH, and in children | 7 months
  Proportion of participants with AESIs throughout the study period

SECONDARY OUTCOMES:
To determine binding LASV-GPC-specific antibody responses induced by rVSV∆G-LASV-GPC vaccine | 6 months/2.5 years
  Proportion of participants with binding antibody responses to LASV-GPC
To determine binding LASV-GPC-specific antibody responses induced by rVSV∆G-LASV-GPC vaccine | 6 months/2.5 years
  Magnitude of binding antibody responses to LASV-GPC
To determine neutralizing LASV-GPC-specific antibody responses induced by rVSV∆G-LASV-GPC vaccine in a subset of participants in each group | 6 months/2.5 years
  Proportion of participants with neutralizing antibody responses against LASV
To determine neutralizing LASV-GPC-specific antibody responses induced by rVSV∆G-LASV-GPC vaccine in a subset of participants in each group | 6 months/2.5 years
  Magnitude of neutralizing antibody responses against LASV
To evaluate the magnitude and duration of the rVSV∆G-LASV-GPC vaccine viremia in plasma in a subset of participants | 6 months/2.5 years
  Magnitude and duration of rVSV∆G-LASV-GPC vaccine viremia by culture
To evaluate the magnitude and duration of the rVSV∆G-LASV-GPC vaccine viremia in plasma in a subset of participants | 6 months/2.5 years
  Magnitude and duration of rVSV∆G-LASV-GPC vaccine shedding in urine and saliva by culture
To evaluate the magnitude and duration of the rVSV∆G-LASV-GPC vaccine shedding in saliva and urine, and possibly semen and cervicovaginal fluid, in a subset of participants | 6 months/2.5 years
  Magnitude and duration of rVSV∆G-LASV-GPC vaccine shedding in semen and cervicovaginal secretions by culture

CONTACTS AND LOCATIONS:
Locations (3):
- Noguchi Memorial Institute for Medical Research (NMIMR), Accra, Ghana
- PREVAIL_ John F. Kennedy Medical Center (JFK), Monrovia, Liberia
- Walter Reed Program - Nigeria, Wuse, Nigeria

IPD SHARING:
Plan to Share IPD: No